CLINICAL TRIAL: NCT07204860
Title: menuCH-Kids, the First Swiss National Nutrition Survey in Children and Adolescents
Acronym: menuCH-Kids
Status: Completed | Type: Observational
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Federal Food Safety and Veterinary Office (Unknown); Berner Fachhochule (Unknown); Kinderklinik Inselspital (Unknown); Università della Svizzera italiana (Unknown); Ospedale Regionale di Bellinzona (Unknown); Universität Zürich (Unknown); Ostschweizer Kinderspital (Other); Kinderspital Luzern (Unknown); Zürcher Hochschule für Angewandte Wissenschaften (Unknown); Haute école spécialisée de Suisse occidentale (Unknown); Swiss Nutrition and Health Foundation (Unknown); YouGov Schweiz (Unknown)
Responsible Party: Sponsor
Other Study IDs: menuCH-Kids_2022-01602
Record Dates: First submitted 2025-08-18; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Nutrition Assessment; Healthy Adolescents; Healthy Children; Population Study; Random Sample; Switzerland; Diet Habits; Biomarkers
Keywords: children; adolescents; nutrition biomarkers; 24HDRs; Swiss; populational nutrition survey; dietary assessement; diet
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood and urine samples, analysed for nutritional status, health status and contaminents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Public health study on the nutritional status and eating habits of children and adolescents in Switzerland

DETAILED DESCRIPTION:
This multicentric descriptive cross-sectional observational study, including randomly selected children from 6 to 17 years old living in six regions of Switzerland (Vaud, Bern, Zurich, Luzern, St Gallen, Ticino), provide valuable information on the nutritional status of Swiss children.

The aims of this study were to 1) characterize the diet and health behaviors of children and adolescents (who eats what, how much, when, where and with whom); 2) determine the nutritional status, energy and macro- and micro-nutrient intake of children and adolescents; 3) estimate the daily intake of contaminants and other harmful substances; 4) derive population-based national reference values for selected micronutrients and vitamins.

It collected high quality representative data on food consumption, dietary and health behaviours (two 24h recalls, which are extensive interviews qualitative and quantitative about the diet of the previous day, and an online questionnaire on food propensity and dietary habits, lifestyle and sociodemographic data) as well as anthropometric and body composition parameters, blood pressure and biological samples (urine spot, optional venous blood).

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free-living children aged between 6 and 17 years
* Permanent residents in Switzerland
* Participants and their legal guardian(s) must be able to read and speak German, French or Italian
* Informed consent provided

Exclusion Criteria:

* Known severe chronic disease (e.g. renal, gastrointestinal, cognitive disorder)
* Hospitalization (overnight stay in the last four weeks before the visit)
* Pregnancy and breastfeeding
* Insufficient knowledge of German, French or Italian or inability to understand the study and/or to provide informed consent
* Inability to come to recruitment center
* Refusal to be informed about study incidental findings concerning the child

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Invited individuals were randomly selected from the Swiss cantonal population registries using the Federal Statistical Office (FSO) sampling frame. The sample of invited persons consisted in 6-17yo children and adolescents residing in Swiss municipalities located within a 30 minutes travel-time to the 6 investigation centers (Bellinzona, Bern, Lausanne, Luzern, St. Gallen, Zurich), stratified in three age groups : 6-9yo, 10-13yo, 14-17yo
Sampling Method: Probability Sample
Enrollment: 1852 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Dietary intake | baseline
  Dietary intake was captured using two 24-hours recalls using GloboDiet, a multi-pass semi-automatic software, as well as a short food propensity questionaire (FPQ).
Nutritional biomarkers | baseline
  Several nutritional biomarkers will be measured in urine and blood, including blood formula, glycated heamoglobin, lipids (cholesterol types, triglycerides), vitamins (D, B9, B12, beta-caroten), ferritin, calcium. More anaylsis will be performed as the biobanked samples will be analysed, a complete updated list will be available on the study data repository.
physical measurements | baseline
  weight (kg), height (cm), blood pressure (mmHg), waist and hip circumference (cm)
Lifestyle | baseline
  A questionnaire containing lifestyle information, including physical activity, screentime, sleep, eating and cooking habits, dietary supplements, health status. The full questionnaire content is available on the data repository website.
socio-demographic information | baseline
  The questionnaire include information about the household, including parent's education and job type, household size, nationality etc. We also have information from the Federal Office of statistics, including typology of their adress (urban vs rural), a spatial socioeconomic proxy (Swiss-SEP), sex and age of the participant... A complete list is available on the study data repository.

CONTACTS AND LOCATIONS:
Locations (6):
- Switzerland (6):
  - Ospedale Regionale di Bellinzona, Istituto Pediatrico della Svizzera Italiana, Bellinzona
  - Kinderklinik Inselspital, Bern
  - Unisante, Lausanne
  - Kinderspital Luzern (LUKS), Lucerne
  - Ostschweizer Kinderspital (OKS), Sankt Gallen
  - Universität Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
All data will be accessible in a data repository from the Federal Food Safety and Veterinary Office, who mandeted and financed the study
Time Frame: It will be available from Autumn 2025
Access Criteria: Data will be accessible to researchers, after signing a data protection agreement. Access to licensed datasets will only be granted when the Lead Researcher is an employee of a legally registered receiving agency (university, research company, research centre, national or international research organization, etc.) on behalf of which access to the data is requested. Commercial use of the data is not permitted. The Lead Researcher assumes all responsibility for compliance with all terms of this Data Access Agreement by all researchers involved in the respective research project.
URL: https://www.studydata.blv.admin.ch/home

REFERENCES:
- See also: website of the stuy. Results, data access links and other information can be found there — http://menuch-kids.ch